CLINICAL TRIAL: NCT01000506
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Dose Ranging Study to Determine the Effect of Mepolizumab on Exacerbation Rates in Subjects With Severe Uncontrolled Refractory Asthma
Brief Title: Dose Ranging Efficacy And Safety With Mepolizumab in Severe Asthma
Acronym: DREAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112997
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: Dose-ranging; Safety; Pharmacodynamics; eosinophils; SB-240563; Efficacy; Severe refractory asthma; mepolizumab; Placebo
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mepolizumab 750mg (Active Comparator): Mepolizumab 750mcg i.v. every 4 weeks
  Interventions: Biological: Mepolizumab 750
- Mepolizumab 250mg (Active Comparator): Mepolizumab 250mcg i.v. every 4 weeks
  Interventions: Biological: Mepolizumab 250
- Mepolizumab 75mg (Active Comparator): Mepolizumab 75mcg i.v. every 4 weeks
  Interventions: Biological: Mepolizumab 75
- Placebo (Placebo Comparator): Placebo saline every 4 weeks i.v.
  Interventions: Drug: Placebo saline

INTERVENTIONS:
Biological: Mepolizumab 750 — Mepolizumab 750mg every four weeks by i.v.
  Arms: Mepolizumab 750mg
Biological: Mepolizumab 250 — Mepolizumab 250mg every four weeks by i.v.
  Arms: Mepolizumab 250mg
Biological: Mepolizumab 75 — Mepolizumab 75mg every four weeks by i.v.
  Arms: Mepolizumab 75mg
Drug: Placebo saline — Placebo saline every four weeks by i.v.
  Arms: Placebo

SUMMARY:
The purpose of this study is to show whether mepolizumab given every 4 weeks intravenously (i.v.) can reduce the frequency of asthma exacerbations in subjects with severe asthma despite receiving high doses of standard asthma medications. The study will look at different doses of mepolizumab in comparison to a placebo.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled study to evaluate the efficacy, safety and pharmacodynamics of three doses (75 mg, 250 mg and 750 mg) of mepolizumab intravenous (i.v.) administered every 4 weeks compared with placebo over a 52-week treatment period in subjects with severe uncontrolled refractory asthma. Efficacy will be measured by the frequency of asthma exacerbations. In addition lung function, rescue medication usage, daily symptoms, asthma control score, asthma quality of life score and withdrawals due to asthma exacerbations will be assessed. Safety will be assessed by adverse events, clinical laboratory evaluations, ECGs, immunogenicity and vital signs. Pharmacodynamics will be assessed by eosinophil levels in blood, serum IL-5 and eosinophil levels in induced sputum.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 12 to 65 years inclusive
* Minimum weight 45kg
* Clinical features of severe refractory asthma
* Well documented requirement for high dose inhaled corticosteroids (ICS) [i.e. >= 880mcg/day fluticasone propionate or equivalent daily] for at least 12 months
* Using additional controller medication in addition to high dose ICS for at least 12 months
* Persistent airflow obstruction indicated by a pre-bronchodilator FEV1<80% predicted at visit 1 or 2 or peak flow diurnal variability of >20% on 3 or more days during the run-in
* Airway inflammation which is likely to be eosinophilic in nature demonstrated by either raised peripheral blood eosinophils (>=300/microL), sputum eosinophils (>=3%), exhaled nitric oxide (>=50ppb) or prompt deterioration of asthma control following a <=25% reduction in regular maintenance dose of inhaled or oral corticosteroids (OCS)
* History of 2 or more exacerbations requiring systemic corticosteroids in the previous 12 months
* Evidence of asthma documented by airway reversibility, airway hyperresponsiveness or airflow variability
* ECG assessment demonstrating QTc<450msec or QTc<480msec for patients with bundle branch block
* Liver function tests demonstrating ALT<2xUpper Limit of Normal (ULN), AST<2xULN, Alk Phos <=1.5xULN, bilirubin <=1.5xULN
* Female of non-child-bearing potential or child-bearing potential with a negative pregnancy test at screening and prepared to agree to an acceptable method of contraception
* Able to give written informed consent
* Able to read, comprehend and write at a sufficient level to complete study materials

Exclusion Criteria:

* Current smokers or smoking history of >=10 pack years
* Clinically important lung condition other than asthma
* Diagnosis of malignancy or in the process of investigation
* Unstable liver disease
* Churg-Strauss syndrome
* Using methotrexate, troleandomycin, oral gold, cyclosporine, azathioprine or any experimental anti-inflammatory therapy within 3 months of screening
* Omalizumab (Xolair) or any other biological for the treatment of inflammatory disease within 6 months of Visit 1
* Regular use of oral or systemic corticosteroids for diseases other than asthma within 12 months or any intra-articular, short-acting intramuscular corticosteroid within 1 month or intramuscular, long-acting depot corticosteroid within 3 months
* Allergy/intolerance to the excipients in the mepolizumab formulation
* Any investigational drug within 30 days or 5 terminal half-lives, whichever is longer
* Pregnant or breastfeeding or planning to become pregnant
* Clinically significant disease which is uncontrolled with standard treatment
* History of alcohol misuse or substance abuse
* Parasitic infestation within previous 6 months
* Known immunodeficiency
* Unable to follow instructions, use the electronic diary or peak flow meter
* Known evidence of lack of adherence to controller medications and/or follow physician's recommendations
* Previous participation in a study of mepolizumab and received study medication within 90 days

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2009-11-01; Primary Completion 2012-03-23 (Actual); Study Completion 2012-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- United States (21):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Madison, Wisconsin
- Argentina (4):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Québec, Quebec
- Chile (4):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Talcahuano
- France (5):
  - GSK Investigational Site, Clamart
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Saint-Pierre
- Germany (6):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zawadzkie
  - GSK Investigational Site, Zgierz
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Târgu Mureş
- Russia (6):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
- South Korea (4):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Ukraine (7):
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
- United Kingdom (4):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Derived] Chen W, Reddel HK, FitzGerald JM, Beasley R, Janson C, Sadatsafavi M. Can we predict who will benefit most from biologics in severe asthma? A post-hoc analysis of two phase 3 trials. Respir Res. 2023 May 2;24(1):120. doi: 10.1186/s12931-023-02409-2. PMID 37131185
- [Derived] Gibson PG, Prazma CM, Chupp GL, Bradford ES, Forshag M, Mallett SA, Yancey SW, Smith SG, Bel EH. Mepolizumab improves clinical outcomes in patients with severe asthma and comorbid conditions. Respir Res. 2021 Jun 7;22(1):171. doi: 10.1186/s12931-021-01746-4. PMID 34098955
- [Derived] Kim MK, Park HS, Park CS, Min SJ, Albers FC, Yancey SW, Mayer B, Kwon N. Efficacy and safety of mepolizumab in Korean patients with severe eosinophilic asthma from the DREAM and MENSA studies. Korean J Intern Med. 2021 Mar;36(2):362-370. doi: 10.3904/kjim.2019.198. Epub 2020 May 26. PMID 32450626
- [Derived] Ortega HG, Meyer E, Brusselle G, Asano K, Prazma CM, Albers FC, Mallett SA, Yancey SW, Gleich GJ. Update on immunogenicity in severe asthma: Experience with mepolizumab. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2469-2475.e1. doi: 10.1016/j.jaip.2019.03.042. Epub 2019 Apr 5. No abstract available. PMID 30954640
- [Derived] Ortega H, Yancey SW, Keene ON, Gunsoy NB, Albers FC, Howarth PH. Asthma Exacerbations Associated with Lung Function Decline in Patients with Severe Eosinophilic Asthma. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):980-986.e1. doi: 10.1016/j.jaip.2017.12.019. Epub 2018 Feb 15. PMID 29398640
- [Derived] Gunsoy NB, Cockle SM, Yancey SW, Keene ON, Bradford ES, Albers FC, Pavord ID. Evaluation of Potential Continuation Rules for Mepolizumab Treatment of Severe Eosinophilic Asthma. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):874-882.e4. doi: 10.1016/j.jaip.2017.11.026. Epub 2017 Dec 16. PMID 29258789
- [Derived] Ortega H, Li H, Suruki R, Albers F, Gordon D, Yancey S. Cluster analysis and characterization of response to mepolizumab. A step closer to personalized medicine for patients with severe asthma. Ann Am Thorac Soc. 2014 Sep;11(7):1011-7. doi: 10.1513/AnnalsATS.201312-454OC. PMID 24983709
- [Derived] Prazma CM, Wenzel S, Barnes N, Douglass JA, Hartley BF, Ortega H. Characterisation of an OCS-dependent severe asthma population treated with mepolizumab. Thorax. 2014 Dec;69(12):1141-2. doi: 10.1136/thoraxjnl-2014-205581. Epub 2014 May 16. PMID 24834924
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112997 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) who met the eligibility criteria at screening, entered the two week Run-in phase and par. who met the randomization eligibility criteria at the end of the Run-in phase entered into the 52-week Double-blind treatment period followed by a 4-week Follow-up phase. The total duration of participation in the study was 58 Weeks.
Pre-assignment Details: A total of 888 par. were enrolled, of these, 168 were screen failures and 720 entered the run-in phase. 99 participants were run-in failures and 621 completed the run-in phase and were randomized. Of these, 616 participants were randomized and received treatment and were included within the Intent-to-Treat (ITT) Population.
Groups:
- Placebo IV: Participants received placebo intravenous (IV) infusion every 4 weeks for 48 weeks (giving 52 weeks of exposure to investigational product).
- Mepolizumab 75 mg IV: Participants received mepolizumab 75 milligrams (mg) IV infusion every 4 weeks for 48 weeks (giving 52 weeks of exposure to investigational product).
- Mepolizumab 250 mg IV: Participants received mepolizumab 250 mg IV infusion every 4 weeks for 48 weeks (giving 52 weeks of exposure to investigational product).
- Mepolizumab 750 mg IV: Participants received mepolizumab 750 mg IV infusion every 4 weeks for 48 weeks (giving 52 weeks of exposure to investigational product).
Period: Overall Study
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Started | 155 | 153 | 152 | 156
Completed | 127 | 129 | 131 | 133
Not Completed | 28 | 24 | 21 | 23
Not completed — Adverse Event | 6 | 5 | 8 | 9
Not completed — Lack of Efficacy | 8 | 6 | 4 | 4
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 4 | 0
Not completed — Physician Decision | 1 | 3 | 3 | 3
Not completed — Withdrawal by Subject | 11 | 8 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Mepolizumab 75 mg IV: Participants received mepolizumab 75 mg IV infusion every 4 weeks for 48 weeks (giving 52 weeks of exposure to investigational product).
- Total: Total of all reporting groups
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV | Total
Number analyzed (Participants) | 155 | 153 | 152 | 156 | 616
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (11.33) | 50.2 (10.84) | 49.4 (11.63) | 48.6 (11.06) | 48.6 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 104 | 93 | 93 | 387
  Male | 58 | 49 | 59 | 63 | 229
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6 | 5 | 8 | 5 | 24
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 1 | 2 | 0 | 2 | 5
  Asian - East Asian Heritage | 7 | 6 | 7 | 6 | 26
  Asian - South East Asian Heritage | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White - Arabic/North African Heritage | 3 | 1 | 2 | 1 | 7
  White - White/Caucasian/European Heritage | 137 | 138 | 133 | 139 | 547
  Mixed Race | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Significant Exacerbations of Asthma Per Year
Description: Clinically significant exacerbations of asthma are defined as worsening of asthma which required use of oral/systemic corticosteroids (for participants on maintenance oral corticosteroids [OCS], an exacerbation requiring OCS is defined as the use of oral/systemic corticosteroids at least double the existing maintenance dose for at least 3 days) and/or hospitalization and/or emergency department (ED) visit. The frequency of clinically significant exacerbations of asthma over the 52-week treatment period is expressed as exacerbation rate per year. Analysis of the number of exacerbations was performed using a negative binomial regression model with covariates of treatment group, Baseline (BL) maintenance OCS therapy (OCS vs. no OCS), region, exacerbations in the year prior to the study (as an ordinal variable) and BL percent (%) predicted forced expiratory volume in 1 second (FEV1), and with logarithm of time on treatment as an offset variable
Time Frame: From randomization (Week 0) to Week 52 or early withdrawal (EW)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and who received at least one dose of study medication.
Measure: Number; unit: Exacerbations per year
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Exacerbations per year | 2.40 | 1.24 | 1.46 | 1.15
Statistical Analysis 1: Comparison: Placebo IV vs Mepolizumab 75 mg IV; Test type: Superiority or Other; p < 0.001, Negative Binomial regression model — Hochberg testing procedure with a one-sided alpha of 2.5% used for controlling multiplicity; Rate Ratio = 0.52, 95% CI 2-sided [0.39 to 0.69] — Number of exacerbations per year in the mepolizumab 75mg IV arm divided by the number of exacerbations per year in the placebo arm
Statistical Analysis 2: Comparison: Placebo IV vs Mepolizumab 250 mg IV; Test type: Superiority or Other; p < 0.001, Negative Binomial regression model — Hochberg testing procedure with a one-sided alpha of 2.5% used for controlling multiplicity; Rate Ratio = 0.61, 95% CI 2-sided [0.46 to 0.81] — Number of exacerbations per year in the mepolizumab 250 mg IV arm divided by the number of exacerbations per year in the placebo arm
Statistical Analysis 3: Comparison: Placebo IV vs Mepolizumab 750 mg IV; Test type: Superiority or Other; p < 0.001, Negative Binomial regression model — Hochberg testing procedure with a one-sided alpha of 2.5% used for controlling multiplicity; Rate Ratio = 0.48, 95% CI 2-sided [0.36 to 0.64] — Number of exacerbations per year in the mepolizumab 750 mg IV arm divided by the number of exacerbations per year in the placebo arm

2. Secondary Outcome: Time to First Clinically Significant Exacerbation Requiring Oral or Systemic Corticosteroid, Hospitalization and/ or ED Visit
Description: Clinically significant exacerbations of asthma are defined as worsening of asthma which required use of oral/systemic corticosteroids (for participants on maintenance OCS, an exacerbation requiring OCS is defined as the use of oral/systemic corticosteroids at least double the existing maintenance dose for at least 3 days) and/or hospitalization and/or ED visit. Kaplan-Meier estimates of the probability of an exacerbation is expressed as percentage of participants with an exacerbation over time (by Week 16, Week 32 and Week 52).
Time Frame: From randomization (Week 0) to Week 52 or EW
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Percentage of participants
  Week 16 | 45.2 [37.7 to 53.5] | 22.8 [16.8 to 30.4] | 26.8 [20.4 to 34.7] | 18.9 [13.5 to 26.1]
  Week 32 | 60.4 [52.6 to 68.2] | 38.2 [30.9 to 46.7] | 45.5 [37.9 to 53.9] | 39.9 [32.4 to 48.3]
  Week 52 | 69.7 [62.1 to 77.0] | 48.5 [40.6 to 57.0] | 58.3 [50.4 to 66.4] | 50.1 [42.2 to 58.6]

3. Secondary Outcome: Number of Exacerbations Requiring Hospitalization (Including Intubation and Admittance to an Intensive Care Unit [ICU]) or ED Visit Per Year
Description: The frequency of exacerbations of asthma requiring hospitalization (including intubation and admittance to an intensive care unit [ICU]) or ED visit over the 52-week treatment period is expressed as exacerbation rate per year. Analysis of the number of exacerbations was performed using a negative binomial regression model with covariates of treatment group, Baseline (BL) maintenance OCS therapy (OCS vs. no OCS), region, exacerbations in the year prior to the study (as an ordinal variable) and BL percent (%) predicted forced expiratory volume in 1 second (FEV1), and with logarithm of time on treatment as an offset variable.
Time Frame: From randomization (Week 0) to Week 52 or EW
Population: ITT Population
Measure: Number; unit: Exacerbations per year
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Exacerbations per year | 0.43 | 0.17 | 0.25 | 0.22

4. Secondary Outcome: Time to First Exacerbation Requiring Hospitalization or ED Visit
Description: Exacerbations of asthma requiring hospitalization or ED visit were assessed. Kaplan-Meier estimates of the probability of an exacerbation is expressed as percentage of participants with an exacerbation over time (by Week 16, Week 32 and Week 52).
Time Frame: From randomization (Week 0) to Week 52 or EW
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Percentage of participants
  Week 16 | 8.6 [5.1 to 14.3] | 3.4 [1.4 to 7.9] | 6.7 [3.6 to 12.0] | 3.9 [1.8 to 8.5]
  Week 32 | 14.8 [10.0 to 21.6] | 8.3 [4.8 to 14.1] | 15.1 [10.2 to 22.1] | 8.0 [4.6 to 13.7]
  Week 52 | 18.5 [13.0 to 25.8] | 10.4 [6.4 to 16.7] | 15.9 [10.8 to 22.9] | 12.4 [8.0 to 18.9]

5. Secondary Outcome: Number of All Recorded Exacerbations Per Year
Description: Clinically significant exacerbations (ex) of asthma are defined as worsening of asthma which required use of oral/systemic corticosteroids (for par. on maintenance OCS, an ex requiring OCS is defined as the use of oral/systemic corticosteroids at least double the existing maintenance dose for at least 3 days) and/or hospitalization and/or ED visit. In the case, an event described as an ex was not associated with a deterioration in >=1 of the objectives of eDiary parameters, the investigator (inv) provided an explanation to support the decision for defining the event as an ex. All recorded ex were defined as those recorded by inv, regardless of the outcome of the ex review process. Analysis was performed using Negative Binomial regression model with covariates of treatment group, BL maintenance OCS therapy (OCS vs. no OCS), region, ex in the year prior to the study (as an ordinal variable) and BL % predicted FEV1, and with logarithm of time on treatment as an offset variable.
Time Frame: From randomization (Week 0) to Week 52 or EW
Population: ITT Population
Measure: Number; unit: Exacerbations per year
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Exacerbations per year | 2.46 | 1.34 | 1.49 | 1.20

6. Secondary Outcome: Time to First All Recorded Exacerbation
Description: All recorded exacerbations are defined as those recorded by investigators, regardless of the outcome of the exacerbation review process. In the case, an event described as an exacerbation was not associated with a deterioration in at least one of the objectives of eDiary parameters, the investigator provided an explanation to support the decision for defining the event as an exacerbation. Kaplan-Meier estimates of the probability of an exacerbation is expressed as percentage of participants with an exacerbation over time (by week 16, week 32 and week 52).
Time Frame: From randomization (Week 0) to Week 52 or EW
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Percentage of participants
  Week 16 | 45.9 [38.3 to 54.1] | 26.1 [19.8 to 33.9] | 27.5 [21.0 to 35.4] | 19.6 [14.1 to 26.8]
  Week 32 | 60.9 [53.2 to 68.8] | 41.5 [34.0 to 49.9] | 45.5 [37.8 to 53.9] | 40.5 [33.1 to 48.9]
  Week 52 | 70.1 [62.6 to 77.3] | 52.2 [44.3 to 60.6] | 58.3 [50.4 to 66.4] | 50.8 [42.9 to 59.2]

7. Secondary Outcome: Mean Change From Baseline in Clinic Pre-bronchodilator FEV1 Over the 52-week Treatment Period
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry at each clinic visit. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and the Baseline value. Analysis was performed using mixed model repeated measures with covariates of Baseline, region, Baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), treatment and visit, plus interaction terms for visit by Baseline and visit by treatment group.
Time Frame: From Baseline up to Week 52 or EW
Population: ITT Population. Only those participants available at the specified time points were analyzed for each treatment and represented as n=X, X, X, X respectively.
Measure: Least Squares Mean (Standard Error); unit: Milliliters (mL)
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Milliliters (mL)
  Week 4, n=154, 151, 151, 155 | 149 (35.3) | 163 (35.6) | 137 (35.3) | 112 (34.9)
  Week 8, n=152, 149, 149, 154 | 154 (36.0) | 165 (36.3) | 133 (36.1) | 142 (35.6)
  Week 12, n=150, 147, 148, 151 | 118 (36.5) | 129 (36.9) | 115 (36.5) | 136 (36.1)
  Week 16, n=143, 147, 144, 150 | 135 (37.4) | 137 (37.4) | 97 (37.3) | 94 (36.7)
  Week 20, n=141, 144, 142, 147 | 131 (37.3) | 155 (37.3) | 89 (37.1) | 124 (36.6)
  Week 24, n=136, 138, 141, 141 | 148 (38.7) | 153 (38.7) | 148 (38.3) | 123 (38.0)
  Week 28, n=135, 136, 139, 141 | 125 (37.9) | 176 (37.9) | 89 (37.5) | 95 (37.1)
  Week 32, n=134, 136, 139, 137 | 139 (37.6) | 142 (37.6) | 134 (37.2) | 43 (37.0)
  Week 36, n=132, 136, 137, 135 | 88 (36.7) | 138 (36.6) | 133 (36.3) | 119 (36.1)
  Week 40, n=129, 133, 135, 135 | 125 (38.9) | 180 (38.8) | 140 (38.4) | 87 (38.1)
  Week 44, n=127, 133, 134, 134 | 125 (37.4) | 153 (37.1) | 93 (36.8) | 111 (36.6)
  Week 48, n=128, 132, 133, 133 | 91 (36.7) | 140 (36.5) | 123 (36.2) | 112 (36.0)
  Week 52, n=127, 129, 129, 132 | 60 (37.7) | 121 (37.6) | 140 (37.3) | 115 (36.9)

8. Secondary Outcome: Mean Change From Baseline in Clinic Post-bronchodilator FEV1 Over the 52-week Treatment Period
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in 1 second. Post-bronchodilator FEV1 measurements were taken by spirometry at Baseline, Week 16, Week 32 and Week 52. Post bronchodilator values were recorded following reversibility testing, using the maximum post bronchodilator method. Participants unable to achieve >=12% reversibility and 200 mL change at Visit 1, reversibility test was repeated at Visit 2. These procedures to achieve the maximum post-bronchodilator are generated by the Asthma Clinical Research Network. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and the Baseline value. Analysis was performed using mixed model repeated measures with covariates of Baseline, region, Baseline maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), treatment and visit, plus interaction terms for visit by Baseline and visit by treatment
Time Frame: From Baseline up to Week 52 or EW
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
mL
  Week 16, n=142, 140, 141, 147 | 59 (37.6) | 77 (37.5) | 50 (37.3) | 87 (36.3)
  Week 32, n=130, 132, 133, 132 | 40 (37.8) | 49 (37.5) | 72 (37.2) | 17 (36.8)
  Week 52, n=126, 128, 129, 130 | -9 (36.7) | 36 (36.4) | 80 (36.1) | 69 (35.6)

9. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire (ACQ) Score Over the 52-week Treatment Period
Description: The ACQ-6 is a six-item questionnaire. The six questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, shortness of breath, wheeze) and use of short-acting bronchodilator over the previous week. The response options for all these questions consist of a 0 (no impairment/limitation) to 6 (total impairment/ limitation) scale. The overall ACQ score is calculated as the mean of the 6 questions and therefore ranges between 0 (totally controlled) and 6 (severely uncontrolled). Change from BL is defined as the difference between the value of the endpoint at the time point of interest and BL value. Analysis was performed using mixed model repeated measures with covariates of BL, region, BL maintenance OCS therapy (OCS vs. no OCS), exacerbations in the year prior to the study (as an ordinal variable), BL % predicted FEV1, treatment and visit, plus interaction terms for visit by BL and visit by treatment group.
Time Frame: From Baseline up to Week 52 or EW
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Number analyzed (Participants) | 155 | 153 | 152 | 156
Scores on a scale
  Week 4, n=146, 139, 148, 150 | -0.45 (0.076) | -0.61 (0.077) | -0.50 (0.075) | -0.56 (0.075)
  Week 8, n=147, 140, 142, 145 | -0.50 (0.080) | -0.73 (0.081) | -0.60 (0.080) | -0.65 (0.079)
  Week 12, n=148, 142, 144, 147 | -0.63 (0.080) | -0.79 (0.081) | -0.65 (0.080) | -0.72 (0.079)
  Week 16, n=138, 143, 143, 146 | -0.59 (0.085) | -0.80 (0.085) | -0.52 (0.084) | -0.76 (0.083)
  Week 20, n=138, 140, 137, 139 | -0.59 (0.081) | -0.82 (0.081) | -0.61 (0.080) | -0.72 (0.080)
  Week 24, n=135, 133, 138, 137 | -0.66 (0.080) | -0.85 (0.080) | -0.70 (0.079) | -0.79 (0.079)
  Week 28, n=131, 135, 135, 136 | -0.70 (0.082) | -0.81 (0.081) | -0.66 (0.080) | -0.73 (0.080)
  Week 32, n=130, 133, 136, 136 | -0.62 (0.084) | -0.74 (0.084) | -0.76 (0.083) | -0.74 (0.083)
  Week 36, n=129, 133, 133, 134 | -0.60 (0.082) | -0.78 (0.082) | -0.75 (0.081) | -0.76 (0.081)
  Week 40, n=126, 128, 129, 131 | -0.64 (0.090) | -0.76 (0.090) | -0.73 (0.089) | -0.67 (0.089)
  Week 44, n=123, 125, 129, 129 | -0.62 (0.089) | -0.75 (0.089) | -0.77 (0.087) | -0.69 (0.087)
  Week 48, n=122, 130, 130, 129 | -0.63 (0.085) | -0.72 (0.084) | -0.74 (0.083) | -0.68 (0.084)
  Week 52, n=121, 127, 126, 129 | -0.59 (0.087) | -0.75 (0.087) | -0.87 (0.086) | -0.80 (0.086)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were defined as events occurring from the first dose of investigational product until 4 weeks after the last dose of investigational product, up to 52 weeks.
Description: SAEs and Non-serious AEs were collected for participants of safety population identical to the ITT population, comprised of all participants who were randomized to treatment and who received at least one dose of study medication.
Arm/Group | Placebo IV | Mepolizumab 75 mg IV | Mepolizumab 250 mg IV | Mepolizumab 750 mg IV
Serious Adverse Events (participants affected / at risk) | 25/155 | 20/153 | 24/152 | 19/156
Other Adverse Events (participants affected / at risk) | 106/155 | 113/153 | 113/152 | 112/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=155) | Mepolizumab 75 mg IV (N=153) | Mepolizumab 250 mg IV (N=152) | Mepolizumab 750 mg IV (N=156)
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 16 | 9
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Distributive shock (Vascular disorders) | 0 | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Microlithiasis (General disorders) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Reticulocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=155) | Mepolizumab 75 mg IV (N=153) | Mepolizumab 250 mg IV (N=152) | Mepolizumab 750 mg IV (N=156)
Nasopharyngitis (Infections and infestations) | 24 | 34 | 33 | 29
Upper respiratory tract infection (Infections and infestations) | 15 | 10 | 17 | 19
Bronchitis (Infections and infestations) | 15 | 16 | 13 | 13
Sinusitis (Infections and infestations) | 16 | 10 | 10 | 12
Influenza (Infections and infestations) | 8 | 6 | 5 | 9
Urinary tract infection (Infections and infestations) | 4 | 8 | 8 | 1
Respiratory tract infection (Infections and infestations) | 4 | 4 | 6 | 6
Rhinitis (Infections and infestations) | 7 | 4 | 5 | 3
Lower respiratory tract infection (Infections and infestations) | 4 | 6 | 4 | 4
Pharyngitis (Infections and infestations) | 4 | 8 | 2 | 3
Viral infection (Infections and infestations) | 3 | 5 | 3 | 6
Respiratory tract infection viral (Infections and infestations) | 3 | 4 | 4 | 4
Ear infection (Infections and infestations) | 3 | 6 | 2 | 2
Acute sinusitis (Infections and infestations) | 4 | 5 | 1 | 2
Gastroenteritis (Infections and infestations) | 3 | 4 | 0 | 4
Cystitis (Infections and infestations) | 2 | 4 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 1 | 4 | 1
Tonsillitis (Infections and infestations) | 4 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 11 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 10 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 12 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 6 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5
Headache (Nervous system disorders) | 27 | 32 | 32 | 32
Dizziness (Nervous system disorders) | 2 | 4 | 3 | 6
Migraine (Nervous system disorders) | 1 | 0 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 7 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6 | 9 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 10 | 8 | 12 | 19
Ligament sprain (Injury, poisoning and procedural complications) | 6 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 2 | 8
Nausea (Gastrointestinal disorders) | 3 | 4 | 5 | 4
Vomiting (Gastrointestinal disorders) | 2 | 4 | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 3 | 4
Toothache (Gastrointestinal disorders) | 0 | 5 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 0 | 3 | 2
Oedema peripheral (General disorders) | 7 | 5 | 6 | 3
Fatigue (General disorders) | 4 | 6 | 7 | 2
Chest pain (General disorders) | 4 | 1 | 7 | 3
Injection site reaction (General disorders) | 5 | 5 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 4 | 2
Asthenia (General disorders) | 0 | 4 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 5 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 2 | 0 | 5
Hypertension (Vascular disorders) | 7 | 6 | 6 | 4
Hypersensitivity (Immune system disorders) | 4 | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.